CLINICAL TRIAL: NCT00394316
Title: Autologous Transplantation of Genetically Modified Cells for the Treatment of X-Linked Chronic Granulomatous Disease
Brief Title: Gene Therapy for Chronic Granulomatous Disease
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 070017; 07-I-0017
Record Dates: First submitted 2006-10-31; First posted 2006-11-01 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2014-04-08

CONDITIONS: Chronic Granulomatous Disease
Keywords: CD34 Stem Cells; Busulfan; Gene Therapy; Immune Reconstitution; Engraftment; Chronic Granulomatous Disease (CGD); Gp91 Phox Deficiency; Peripheral Blood Stem Cells; Bone Marrow Transplantation; Chronic Granulomatous Disease; CGD
MeSH Terms: conditions — Granulomatous Disease, Chronic

INTERVENTIONS:
Drug: Phagocyte Oxidase Subunit Transduced CD34 Hematopoietic Stem Cells

SUMMARY:
X-linked Chronic Granulomatous Disease (CGD) is an inherited disorder caused by an abnormal gene that fails to make the protein known as gp91 phox. This protein is part of a group of proteins that work to create hydrogen peroxide in neutrophils. Neutrophils are a type of white blood cell that helps fight infections. As a result, patients who do not make this gp91 phox frequently develop life-threatening infections. In addition, these neutrophils often act abnormally, resulting in the creation of a granuloma, which is an abnormal collection of cells. These granulomas can then become large enough to block organs, such as the bladder and/or intestines, causing significant problems. Patients are usually treated with antibiotics (often needed for extended periods of time) for the infections caused by CGD, and with corticosteroids for the granulomas. However, these drugs do not cure CGD itself, and can have significant side effects. Thus patients with CGD do not have a normal life expectancy.

The only available cure to date for CGD is Bone Marrow Transplantation (BMT), where the blood-making cells from a specially matched brother or sister donor (allogeneic) or a similarly matched unrelated donor are given to the patient after the patient has undergone some kind of chemotherapy or radiation in preparation for receiving the cells. If the cells from the donor engraft (or survive in the marrow), the patient can be cured; however, there is a risk that the cells may not engraft or that they may later get rejected from the body. Also, the cells from the donor can react against the patient, causing a serious disorder called "Graft Versus Host Disease" (GVHD). Although there are a number of methods used to try to reduce and/or prevent graft rejection and/or GVHD, these complications can still occur even with the newer methods now being developed. The risks of such complications are lower when a brother or sister is used as the donor; however, not all patients (even those with siblings) will have an ideally matched donor. Hence, transplantation, especially when using an unrelated donor, is not always a perfect cure.

Because the gene responsible for making the gp91 phox is known, it is possible to use gene therapy to try to cure this disease. In gene therapy, some of the blood-making cells are taken from the patient using a technique called apheresis. The normal gene is placed into the cells using special viruses called retroviruses. The cells are then able to produce the normal protein. In this trial, the patient will receive a small dose of chemotherapy called busulfan, lower than what is traditionally used in allogeneic BMT, and the newly corrected cells will then be put back into the patient.

Even with the best standard of care, a number of patients with CGD will still die from infection. For those patients who have an unresponsive or progressive infection and do not have a possible sibling donor, their only hope is either a Matched Unrelated Donor (MUD) transplant, which has a high risk of causing death itself, or gene therapy. Hence, we would propose using gene therapy in these patients as this has less risk of causing death, but can still possibly offer a cure. Even if the corrected cells do not remain life long to rid the patients entirely of their disease, as long as they persist for even a few months, they would be able to at least clear the current infection for which the patients are being considered for enrollment in this protocol. Further, they would still be eligible to undergo a matched unrelated donor transplant in the event that gene therapy does not confer any benefit.

DETAILED DESCRIPTION:
X-linked Chronic Granulomatous Disease (CGD) is an inherited disorder caused by an abnormal gene that fails to make the protein known as gp91 phox. This protein is part of a group of proteins that work to create hydrogen peroxide in neutrophils. Neutrophils are a type of white blood cell that helps fight infections. As a result, patients who do not make this gp91 phox frequently develop life-threatening infections. In addition, these neutrophils often act abnormally, resulting in the creation of a granuloma, which is an abnormal collection of cells. These granulomas can then become large enough to block organs, such as the bladder and/or intestines, causing significant problems. Patients are usually treated with antibiotics (often needed for extended periods of time) for the infections caused by CGD, and with corticosteroids for the granulomas. However, these drugs do not cure CGD itself, and can have significant side effects. Thus patients with CGD do not have a normal life expectancy.

The only available cure to date for CGD is Bone Marrow Transplantation (BMT), where the blood-making cells from a specially matched brother or sister donor (allogeneic) or a similarly matched unrelated donor are given to the patient after the patient has undergone some kind of chemotherapy or radiation in preparation for receiving the cells. If the cells from the donor engraft (or survive in the marrow), the patient can be cured; however, there is a risk that the cells may not engraft or that they may later get rejected from the body. Also, the cells from the donor can react against the patient, causing a serious disorder called Graft Versus Host Disease (GVHD). Although there are a number of methods used to try to reduce and/or prevent graft rejection and/or GVHD, these complications can still occur even with the newer methods now being developed. The risks of such complications are lower when a brother or sister is used as the donor; however, not all patients (even those with siblings) will have an ideally matched donor. Hence, transplantation, especially when using an unrelated donor, is not always a perfect cure.

Because the gene responsible for making the gp91 phox is known, it is possible to use gene therapy to try to cure this disease. In gene therapy, some of the blood-making cells are taken from the patient using a technique called apheresis. The normal gene is placed into the cells using special viruses called retroviruses. The cells are then able to produce the normal protein. In this trial, the patient will receive a small dose of chemotherapy called busulfan, lower than what is traditionally used in allogeneic BMT. Then the newly corrected cells will be put back into the patient.

Even with the best standard of care, a number of patients with CGD will still die from infection. For those patients who have an unresponsive or progressive infection and do not have a possible sibling donor, their only hope is either a Matched Unrelated Donor (MUD) transplant, which has a high risk of causing death itself, or gene therapy. Hence, we would propose using gene therapy in these patients as this has less risk of causing death, but can still possibly offer a cure. Even if the corrected cells do not remain lifelong to rid the patients entirely of their disease, as long as they persist for even a few months, they would be able to at least clear the current infection for which the patients are being considered for enrollment in this protocol. Further, they would still be eligible to undergo a matched unrelated donor transplant in the event that gene therapy does not confer any benefit.

ELIGIBILITY:
* INCLUSION CRITERIA:

Have a diagnosis of X-linked CGD (i.e., a gp91-phox gene mutation/defect).

* Have a minimum of 5.0 x10(6) CD34 plus cells per kg body weight (collected and cryopreserved, prior to enrollment) available for transduction.
* Weight greater or equal to 20 kg.
* Unresponsive or incurable infection as defined by either/or:

  * Continued (stable or progressive) infection despite standard antimicrobial therapy

    * Stable and/or does not completely resolve despite a minimum of 2 months of treatment

OR

* Progressive as shown by increase in size or new sites of infection despite therapy for a minimum of two weeks.

  * Multidrug resistant organism as determined by tissue analysis

    * Not have a suitable sibling who is HLA-matched for stem cell or bone marrow donation.
    * Males aged 3-55 years.
    * Must use two approved methods of contraception, such as barrier method (condom) with a spermicidal if sexually active
    * Willingness to remain hospitalized for several weeks
    * Have a primary care physician at home
    * Consent to permit storage of blood and/or other tissues samples
    * Patients with a Grade 3 toxicity due to active infection may enter this trial.

EXCLUSION CRITERIA:

* Weigh less than 20 kg.
* Be hemodynamically unstable or requiring pressor support.
* Require ventilatory assistance with high levels of oxygen.
* Have an HLA-matched suitable sibling for stem cell or bone marrow donation.
* Intolerance to busulfan.
* Failure to use two approved methods of contraception, such as barrier method (such as a condom with a spermicidal).
* Participation in another Gene Therapy clinical trial
* If pre-conditioning and pre-infusion evaluations are found to match a criterion for Grade 4 toxicity as defined in Toxicity Table for grading severity of AEs
* Presence of an anti-GP91 antibody.

When the condition or parameter has returned to the criterion for Grade 3 or less for that condition or parameter twice over an interval of at least 4 weeks prior to the infusion, eligibility may be resumed.<TAB><TAB>

Ages: 3 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2006-10-30; Primary Completion 2014-04-08 (Actual); Study Completion 2014-04-08 (Actual)

PRIMARY OUTCOMES:
Can conditioning with busulfan improve gene therapy outcomes

SECONDARY OUTCOMES:
1) To evaluate further the safety of gene therapy2) To monitor long-term results of gene therapy with conditioning

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth M Kang, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] International Chronic Granulomatous Disease Cooperative Study Group. A controlled trial of interferon gamma to prevent infection in chronic granulomatous disease. N Engl J Med. 1991 Feb 21;324(8):509-16. doi: 10.1056/NEJM199102213240801. PMID 1846940
- [Background] Aiuti A, Slavin S, Aker M, Ficara F, Deola S, Mortellaro A, Morecki S, Andolfi G, Tabucchi A, Carlucci F, Marinello E, Cattaneo F, Vai S, Servida P, Miniero R, Roncarolo MG, Bordignon C. Correction of ADA-SCID by stem cell gene therapy combined with nonmyeloablative conditioning. Science. 2002 Jun 28;296(5577):2410-3. doi: 10.1126/science.1070104. PMID 12089448
- [Background] Cavazzana-Calvo M, Hacein-Bey S, de Saint Basile G, Gross F, Yvon E, Nusbaum P, Selz F, Hue C, Certain S, Casanova JL, Bousso P, Deist FL, Fischer A. Gene therapy of human severe combined immunodeficiency (SCID)-X1 disease. Science. 2000 Apr 28;288(5466):669-72. doi: 10.1126/science.288.5466.669. PMID 10784449
- [Derived] Kang EM, Choi U, Theobald N, Linton G, Long Priel DA, Kuhns D, Malech HL. Retrovirus gene therapy for X-linked chronic granulomatous disease can achieve stable long-term correction of oxidase activity in peripheral blood neutrophils. Blood. 2010 Jan 28;115(4):783-91. doi: 10.1182/blood-2009-05-222760. Epub 2009 Dec 1. PMID 19965657